CLINICAL TRIAL: NCT05005065
Title: A Randomized, Open-label, Multiple Dosing, Cross-over Phase 1 Clinical Trial to Evaluate Pharmacokinetics/Pharmacodynamics and Safety/Tolerability of IN-C005 and IN-A001 After Oral Administration in Healthy Caucasian Subjects
Brief Title: Evaluation of the Pharmacokinetics/Pharmacodynamics and Safety/Tolerability of IN-C005 and IN-A001 in Healthy Caucasians
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IN_BTK_102
Record Dates: First submitted 2021-07-05; First posted 2021-08-13 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2021-08

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, multiple dosing, crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment AB (Experimental): Participants will be randomized to receive IN-C005 Y mg (Treatment A) and IN-A001 Y mg (Treatment B) sequentially in a two-period sequence. There will be a washout period of at least 14 days between Period 1 and Period 2.
  Interventions: Drug: IN-A001 Y mg; Drug: IN-C005 Y mg
- Treatment BA (Experimental): Participants will be randomized to receive IN-A001 Y mg and IN-C005 Y mg sequentially in a two-period sequence. There will be a washout period of at least 14 days between Period 1 and Period 2.
  Interventions: Drug: IN-A001 Y mg; Drug: IN-C005 Y mg
- Treatment CD (Experimental): Participants will be randomized to receive IN-C005 Z mg (Treatment C) and IN-C005 X mg (Treatment D) sequentially in a two-period sequence. There will be a washout period of at least 14 days between Period 1 and Period 2.
  Interventions: Drug: IN-C005 X mg; Drug: IN-C005 Z mg
- Treatment DC (Experimental): Participants will be randomized to receive IN-C005 X mg and IN-C005 Z mg sequentially in a two-period sequence. There will be a washout period of at least 14 days between Period 1 and Period 2.
  Interventions: Drug: IN-C005 X mg; Drug: IN-C005 Z mg

INTERVENTIONS:
Drug: IN-C005 X mg — Oral capsule
  Arms: Treatment CD; Treatment DC
Drug: IN-A001 Y mg — Oral tablet
  Arms: Treatment AB; Treatment BA
Drug: IN-C005 Y mg — Oral capsule
  Arms: Treatment AB; Treatment BA
Drug: IN-C005 Z mg — Oral capsule
  Arms: Treatment CD; Treatment DC

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics/pharmacodynamics and safety/tolerability of IN-C005 and IN-A001 after oral administration in healthy Caucasian subjects.

DETAILED DESCRIPTION:
[Part 1] To evaluate the pharmacokinetic (PK)/pharmacodynamic (PD) profiles and safety/tolerability of 100 mg IN-C005 versus 100 mg IN-A001 after multiple oral dosing in healthy Caucasian subjects

[Part 2] To evaluate the PK/PD profiles and safety/tolerability of 50 mg IN-C005 versus 75 mg IN-C005 after multiple oral dosing in healthy Caucasian subjects

ELIGIBILITY:
Inclusion Criteria:

1. Is healthy Caucasian adult aged 19 to 50 years (inclusive) at the time of signing the informed consent form (ICF) (A Caucasian is defined as a European who was born in Europe, has the duration of residence outside of Europe less than 10 years, and both of whose parents and grandparents are European-born).
2. Has ≥ 18.0 and ≤ 30.0 kg/m2 of body mass index (BMI) with a body weight (BW) ≥ 55.0 kg at screening.
3. Has a negative result in serum Helicobacter pylori IgG antibody test.
4. Decides to participate voluntarily in the study after being fully informed of and understanding the study completely, and provides his/her written informed consent prior to screening procedure.
5. Is eligible for this study in the opinion of the investigator based on the results of physical examination, clinical laboratory tests, interview, etc.

Exclusion Criteria:

1. Has a history or current evidence of clinically significant disorder of hepatic, renal, nervous, respiratory, endocrine, hemato-oncologic, cardiovascular, urinary, and/or psychiatric system.
2. Has a history or current evidence of gastrointestinal disease that may affect the safety and PD assessments for study treatment (e.g., gastrointestinal ulcer, gastritis, gastric cramp, gastroesophageal reflux disease, and Crohn's disease) or a history of gastrointestinal surgery (except for simple appendectomy or herniotomy).
3. Has a history or current evidence of clinically significant hypersensitivity to study drugs or any ingredient of proton pump inhibitors and other drugs (such as aspirin and antibiotics).
4. Has a positive result on serology tests (for hepatitis B, human immunodeficiency virus [HIV], and hepatitis C).
5. Has a blood level of total bilirubin, AST (GOT), or ALT (GPT) > 1.5 X upper limit of normal (ULN) based on screening procedures including repeated ones.
6. Has a calculated eGFR per MDRD equation < 60 mL/min/1.73 m2 based on screening procedures including repeated ones.
7. Has systolic blood pressure (SBP) of < 90 mmHg or > 140 mmHg, diastolic blood pressure (DBP) of < 50 mmHg or > 95 mmHg, or pulse rate (PR) of < 45 beats/min or > 100 beats/min on vital signs as measured in sitting position after taking a rest for at least 5 minutes at screening.
8. Has an anatomical disorder that precludes insertion and maintenance of intragastric pH meter catheter or is expected to be intolerable to insertion of intragastric pH meter catheter.
9. Has a history of drug abuse or has a positive response to drug abuse on urine drug screening test.
10. Has received any prescription drug or herbal medication within 2 weeks of or any over-the-counter (OTC) drug, dietary supplements, or vitamins within 1 week of scheduled first dose or is expected to receive such medication during the study (Note: a subject may participate in the study at the discretion of the investigator provided the subject meets all the other criteria).
11. Has participated and received an investigational agent in another clinical trial or bioequivalence study within 6 months prior to the first dose of study treatment (Note: This is not applied to participation in another part of this study).
12. Has donated whole blood within 2 months prior to the scheduled first dose, or has donated blood components or received transfusion within a month prior to the scheduled first dose.
13. Has excessive caffeine intake (> 5 units/day), continues the use of alcohol (> 21 units/week, 1 unit = 10 g of pure alcohol), or is unable to stop drinking during hospitalization period.
14. Has a positive result for cotinine on urine drug screening test or is unable to stop smoking throughout the study.
15. Is unable to avoid grapefruit-containing foods during the time from 24 hours (hrs) before hospitalization to discharge in Period 1 and Period 2, respectively.
16. Is unable to avoid caffeine-containing foods (e.g., coffee, tea [red tea, green tee, etc.], soda, coffee milk, and nutritive tonic drink) during the time from 24 hrs before hospitalization to discharge Period 1 and Period 2, respectively.
17. For all women of childbearing potential (WOCBP) excluding those on amenorrhea for at least 12 months and those who underwent surgical sterilization (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), has a positive result for pregnancy test (urine hCG) performed prior to the first dose of study treatment or is pregnant or breastfeeding.
18. Is unable to use a medically acceptable contraceptive method throughout the study. Medically acceptable contraceptive methods include:

    * Use of an intrauterine device with a proven birth control failure rate by the subject or subject's spouse (or partner)
    * Use of (male or female) barrier method with spermicide
    * Surgical sterilization (vasectomy, salpingectomy, tubal ligation, hysterectomy) of the subject or subject's spouse (or partner)
19. Is determined ineligible for study participation by the investigator for other reasons such as clinical laboratory abnormalities.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1, Day 22
  PK: Maximum concentration of drug in plasma
AUClast | Day 1, Day 22
  PK: Area under the plasma drug concentration-time curve from 0 to last point of measurable concentration
Cmax,ss | Day 7 and Day 28
  PK: Maximum (peak) steady-state plasma drug concentration during a dosage interval
AUCtau,ss | Day 7 and Day 28
  PK: Area under the plasma drug concentration-time curve for a dosing interval at steady state
Percent duration of pH ≥4 in 24 hrs (duration %) | Day 1, Day 22
  PD: pH parameter
Percent duration of pH ≥4 in 24 hrs (duration %) | Day 7, Day 28
  PD: pH parameter
Change from baseline in percent duration of pH ≥4 in 24 hrs | Day 1, Day 7, Day 22, Day 28
  PD: pH parameter

SECONDARY OUTCOMES:
AUCinf | Day 1, Day 22
  PK: Area under the plasma drug concentration-time curve from time 0 to infinity
Tmax | Day 1, Day 22
  PK: The time of peak concentration
t1/2 | Day 1, Day 22
  PK: Terminal half-life
CL/F | Day 1, Day 22
  PK: Apparent Clearance
Vd/F | Day 1, Day 22
  PK: Apparent volume of distribution after extravascular administration
Tmax,ss | Day 7, Day 28
  PK: Time to reach Cmax
t1/2,ss | Day 7, Day 28
  PK: Apparent first order terminal elimination half-life
Cmin,ss | Day 7, Day 28
  PK: Minimum observed non zero concentration between dose time and dose time + dosing interval, tau
Cavg,ss | Day 7, Day 28
  PK: The average concentration at steady state, calculated as the ratio of AUCtau to the dosing interval, tau
CLss/F | Day 7, Day 28
  PK: The total body clearance at steady state after oral administration
Vd,ss/F | Day 7, Day 28
  PK: Apparent volume of distribution after extravascular administration in steady state
PTF | Day 7, Day 28
  PK: Peak to trough fluctuation
R | Day 7, Day 28
  PK: Accumulation ratio
Percent duration of pH ≥3 in 24 hrs | Day 1, Day 7, Day 22, Day 28
  PD: pH parameter
Change from baseline in percent duration of pH ≥3 in 24 hrs | Day 1, Day 7, Day 22, Day 28
  PD: pH parameter
Percent duration of pH ≥6 in 24 hrs | Day 1, Day 7, Day 22, Day 28
  PD: pH parameter
Change from baseline in percent duration of pH ≥6 in 24 hrs | Day 1, Day 7, Day 22, Day 28
  PD: pH parameter
Mean and median pH in 24 hrs | Day 1, Day 7, Day 22, Day 28
  PD: pH parameter
Change from baseline in mean pH in 24 hrs | Day 1, Day 7, Day 22, Day 28
  PD: pH parameter
Change from baseline in median pH in 24 hrs | Day 1, Day 7, Day 22, Day 28
  PD: pH parameter
AUEGlast | Day 1, Day 7, Day 22, Day 28
  PD(Gastrin): Area under the concentration-time curve of Serum Gastrin from 0 to last point of quantifiable concentration
Gmax | Day 1, Day 7, Day 22, Day 28
  Gastrin: Maximum gastrin level
ΔAUEGlast | Day 1, Day 7, Day 22, Day 28
  PD(Gastrin): Change from baseline in AUEGlast
ΔGmax | Day 1, Day 7, Day 22, Day 28
  PD(Gastrin): Change from baseline in Gmax

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, MD, Ph.D, Principal Investigator — Clinical Pharmacology and Therapeutics, Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul, Jongro Gu
  - Seoul National University Hopsital, Seoul

IPD SHARING:
Plan to Share IPD: No